CLINICAL TRIAL: NCT01885000
Title: Patient-Reported Outcomes of Brimonidine Tartrate 0.5% Gel for Treatment of Severe Facial Erythema of Rosacea
Brief Title: Patient-Reported Outcome Of Facial Erythema (PROOF)
Acronym: PROOF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RD.03.SPR.29107; 2012-005686-12 (EudraCT Number)
Record Dates: First submitted 2013-06-20; First posted 2013-06-24 (Estimated); Results first posted 2017-01-13 (Estimated); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Rosacea; Erythema
MeSH Terms: conditions — Rosacea; Erythema

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Brimonidine tartrate 0.5% gel (Experimental): Participants applied brimonidine tartrate 0.5% gel topically once daily for 8 days.
  Interventions: Drug: Brimonidine tartrate was applied cutaneously once daily for 8 days.
- Vehicle (Placebo Comparator): Participants applied brimonidine tartrate vehicle gel topically once daily for 8 days.
  Interventions: Drug: Brimonidine tartrate vehicle was applied cutaneously once daily for 8 days.

INTERVENTIONS:
Drug: Brimonidine tartrate was applied cutaneously once daily for 8 days.
  Arms: Brimonidine tartrate 0.5% gel
Drug: Brimonidine tartrate vehicle was applied cutaneously once daily for 8 days.
  Arms: Vehicle

SUMMARY:
The purpose of the study is to evaluate the patient-reported outcomes (feedbacks of patients)of a new drug for the treatment of erythema of rosacea (central facial redness). The feedback of patients receiving the active drug will be compared to the feedback of patients receiving the placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects age of 18 years or older
* A clinical diagnosis of facial rosacea
* A Patient Self-Assessment score of 4 (severe) at Baseline prior to the study drug application
* A Clinician's Erythema Assessment (CEA) score of 3 (moderate) or 4 (severe) at Baseline prior to the study drug application

Exclusion Criteria:

* More than 5 facial inflammatory lesions (papules or pustules) of rosacea
* Any uncontrolled chronic or serious disease or medical condition that may either interfere with the interpretation of the clinical trial results, or put the subject at significant risk if the subject participates in the clinical trial as judged by the investigator
* Known or suspected allergies or sensitivities to any component of the study drugs, including the active ingredient brimonidine tartrate (see Investigator's Brochure)
* Female who is pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2013-07-01 (Actual); Primary Completion 2013-11-14 (Actual); Study Completion 2013-11-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- Germany (7):
  - Klinik für Dermatologie, Venerologie und Allergologie, Berlin
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Klinikum der Johann Wolfgang Goethe-Universität, Frankfurt am Main
  - Universitätsklinikum Münster, Klinik für Hautkrankheiten, Münster
  - Universitäts-Hautklinik Eberhard Karls Universität Tübingen, Tübingen
  - CentroDerm Gesellschaft für dermatolgische Forschung mbH (GmbH), Wuppertal
  - Zentrum für Dermatologie, Allergologie und Dermatochirurgie, Wuppertal
- Sweden (2):
  - Capio Citykliniken, Lund
  - Läkarhuset Odenplan, Stockholm
- United Kingdom (5):
  - NHS Tayside, Dundee
  - University Hospitals of Leicester, Leicester
  - Royal Free Hospital, London
  - Whipps Cross University Hospital, London
  - Harrogate District Hospital, Yorkshire

REFERENCES:
- [Derived] Layton AM, Schaller M, Homey B, Hofmann MA, Bewley AP, Lehmann P, Nohlgard C, Sarwer DB, Kerrouche N, Ma YM. Brimonidine gel 0.33% rapidly improves patient-reported outcomes by controlling facial erythema of rosacea: a randomized, double-blind, vehicle-controlled study. J Eur Acad Dermatol Venereol. 2015 Dec;29(12):2405-10. doi: 10.1111/jdv.13305. Epub 2015 Sep 28. PMID 26416154

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at fourteen centers in Germany, Sweden, United Kingdom from 01 July 2013 (first participant visit) to 14 November 2013 (last participant completed).
Pre-assignment Details: A total of 92 participants were randomized, of which 88 participants completed the study.
Period: Overall Study
Arm/Group | Brimonidine Tartrate 0.5% Gel | Vehicle
Started | 48 | 44
Completed | 46 | 42
Not Completed | 2 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population consisted of the entire population enrolled and randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Brimonidine Tartrate 0.5% Gel | Vehicle | Total
Number analyzed (Participants) | 48 | 44 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (12.9) | 54.9 (12.8) | 54.1 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 26 | 56
  Male | 18 | 18 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 48 | 44 | 92
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Skin phototype [Count of Participants; unit: Participants] — Fitzpatrick skin phototype is a system used to describe a person's skin type. It ranges from skin phototype I to III. Where, skin phototype I = pale white skin, always burns easily, never tans; skin phototype II = fair skin, always burns easily, tans minimally and with difficulty; skin phototype III = darker white skin, burns minimally, tans gradually and uniformly.
  Participants
    Type I | 3 | 6 | 9
    Type II | 34 | 27 | 61
    Type III | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Are Very Satisfied/Satisfied/Somewhat Satisfied With the Overall Study Treatment
Description: Percentage of participants who are very satisfied/satisfied/somewhat satisfied with the study treatment were reported.
Time Frame: Day 8
Population: ITT population consisted of the entire population enrolled and randomized. Here over all number of participants 'N' analyzed signifies number of participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Brimonidine Tartrate 0.5% Gel | Vehicle
Number analyzed (Participants) | 46 | 42
Percentage of participants | 69.6 | 40.4
Statistical Analysis 1: Comparison: Brimonidine Tartrate 0.5% Gel vs Vehicle; Test type: Superiority; p = 0.0065, Cochran-Mantel-Haenszel

2. Primary Outcome: Percentage of Participants With Facial Redness Questionnaire at Day 8
Description: Percentage of participants for each category of facial redness questionnaire on Day 8 was reported. Facial redness questionnaire included 12 questions/categories 1. Satisfied with appearance, 2. Appearance acceptable, 3. Appearance concerned, 4. Embarrassed with facial redness, 5. Self-conscious, 6. Frequency control last 24 hours, 7. Frustrated, 8. Cover up or camouflage, 9. Pay attention to the known triggers, 10. Avoid the known triggers, 11. Interfering with social life, 12. Interfering with work life.
Time Frame: Day 8
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Brimonidine Tartrate 0.5% Gel | Vehicle
Number analyzed (Participants) | 46 | 42
percentage of participants
  1. Very dissatisfied/ Dissatisfied | 45.7 | 69.0
  1. Dissatisfied or Satisfied/Satisfied | 54.3 | 31.0
  2. Very unacceptable/Unacceptable | 47.9 | 59.5
  2.Acceptable or Unacceptable/Acceptable | 52.1 | 40.5
  3.Not at all/Slightly | 28.2 | 21.4
  3. Somewhat /Moderately /Extremely | 71.7 | 78.6
  4. Not at all | 28.3 | 9.5
  4. Slightly/ Somewhat/Moderately/Extremely | 71.7 | 90.4
  5.Not at all/Slightly/ Somewhat: number analyzed (Participants) | 45 | 42
  5.Not at all/Slightly/ Somewhat | 73.4 | 47.6
  5. Moderately/Extremely: number analyzed (Participants) | 45 | 42
  5. Moderately/Extremely | 26.7 | 52.3
  6. Not at all: number analyzed (Participants) | 46 | 41
  6. Not at all | 23.9 | 31.7
  6.Slightly/Somewhat/Moderately/Extremel y: number analyzed (Participants) | 46 | 41
  6.Slightly/Somewhat/Moderately/Extremel y | 76.1 | 68.2
  7. Not at all | 8.7 | 14.3
  7. Slightly/Somewhat/Moderately/Extremely | 91.2 | 85.8
  8.Not at all | 60.9 | 61.9
  8. Slightly/Somewhat | 23.9 | 11.9
  9. Not at all/Rarely: number analyzed (Participants) | 46 | 41
  9. Not at all/Rarely | 47.8 | 48.8
  9.Some of the time/Often/Constantly: number analyzed (Participants) | 46 | 41
  9.Some of the time/Often/Constantly | 52.2 | 51.2
  10.Not at all/Rarely | 47.8 | 47.6
  10. Some of the time/Often/Constantly | 52.2 | 52.4
  11. Not at all | 34.8 | 21.4
  11.Slightly/Somewhat/Moderately/Extremely | 65.2 | 78.5
  12.Not at all: number analyzed (Participants) | 45 | 42
  12.Not at all | 26.7 | 23.8
  12.Slight/Somewhat/Moderate/Extreme/ Not Applicable/I'm not working: number analyzed (Participants) | 45 | 42
  12.Slight/Somewhat/Moderate/Extreme/ Not Applicable/I'm not working | 73.4 | 76.2
Statistical Analysis 1: Comparison: Brimonidine Tartrate 0.5% Gel vs Vehicle; The questionnaire analyzed and reported here is for participants who satisfied with appearance; Test type: Superiority; p = 0.0328, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Brimonidine Tartrate 0.5% Gel vs Vehicle; The questionnaire analyzed and reported here is for participants who appearance acceptable; Test type: Superiority; p = 0.5312, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Brimonidine Tartrate 0.5% Gel vs Vehicle; The questionnaire analyzed and reported here is for participants who appearance concerned; Test type: Superiority; p = 0.0756, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Brimonidine Tartrate 0.5% Gel vs Vehicle; The questionnaire analyzed and reported here is for participants who embarrassed with facial redness; Test type: Superiority; p = 0.0083, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Brimonidine Tartrate 0.5% Gel vs Vehicle; The questionnaire analyzed and reported here is for participants who self-conscious; Test type: Superiority; p = 0.0076, Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: Brimonidine Tartrate 0.5% Gel vs Vehicle; The questionnaire analyzed and reported here is for participants who's frequency control last 24 hours; Test type: Superiority; p = 0.2186, Cochran-Mantel-Haenszel
Statistical Analysis 7: Comparison: Brimonidine Tartrate 0.5% Gel vs Vehicle; The questionnaire analyzed and reported here is for participants who are frustrated; Test type: Superiority; p = 0.2373, Cochran-Mantel-Haenszel
Statistical Analysis 8: Comparison: Brimonidine Tartrate 0.5% Gel vs Vehicle; The questionnaire analyzed and reported here is for participants who cover up or camouflage; Test type: Superiority; p = 0.7769, Cochran-Mantel-Haenszel
Statistical Analysis 9: Comparison: Brimonidine Tartrate 0.5% Gel vs Vehicle; The questionnaire analyzed and reported here is for participants who pay attention to the known triggers; Test type: Superiority; p = 0.8764, Cochran-Mantel-Haenszel
Statistical Analysis 10: Comparison: Brimonidine Tartrate 0.5% Gel vs Vehicle; The questionnaire analyzed and reported here is for participants who avoid the known triggers; Test type: Superiority; p = 0.6149, Cochran-Mantel-Haenszel
Statistical Analysis 11: Comparison: Brimonidine Tartrate 0.5% Gel vs Vehicle; The questionnaire analyzed and reported here is for participants who interfering with social life; Test type: Superiority; p = 0.8361, Cochran-Mantel-Haenszel
Statistical Analysis 12: Comparison: Brimonidine Tartrate 0.5% Gel vs Vehicle; Interfering with work life; Test type: Superiority; p = 0.6259, Cochran-Mantel-Haenszel

3. Primary Outcome: EuroQuality of Life-5 Dimensional-3 Level (EQ-5D-3L) Questionnaire at Day 8
Description: EQ-5D-3L is a 3-level, 5-dimensional format standardized instrument for use as a measure of health outcome used to assess the impact of study treatments on participants quality of life as follows: 1) mobility; 2) self-care; 3) usual activities; 4) pain/discomfort; 5) anxiety/depression. Each dimension comprises 3 levels with corresponding numeric scores, where 1 indicates no problems, and 3 indicates extreme problems. Participant selects answer for each of 5 dimensions considering response that best matches his/her health today with anchors ranging from 0 (worst imaginable health state) to 100 (best imaginable health state). An increase in the EQ-5D-3L total score indicates improvement.
Time Frame: Day 8
Population: ITT population consisted of the entire population enrolled and randomized. Here the over all number of participants analyzed signifies participants who were evaluable for this outcome measure and at specific categories.
Measure: Number; unit: Percentage of participants
Arm/Group | Brimonidine Tartrate 0.5% Gel | Vehicle
Number analyzed (Participants) | 46 | 42
Percentage of participants
  1. I have no problems in walking about | 95.7 | 92.9
  1.I have some problems in walking about | 4.3 | 7.1
  2. I have no problems with self-care | 97.8 | 97.6
  2. I have some problems washing or dressing myself | 2.2 | 2.4
  3.I have no problems with performing usual activity | 91.3 | 90.5
  3.I have some problems with performing usual activity | 8.7 | 9.5
  4.I have no pain or discomfort | 58.7 | 76.2
  4.I have moderate pain or discomfort | 41.3 | 21.4
  4.I have extreme pain or discomfort | 0 | 2.4
  5.I am not anxious or depressed | 87.0 | 73.8
  5.I am moderately anxious or depressed | 10.9 | 26.2
  5.I am extremely anxious or depressed | 2.2 | 0
Statistical Analysis 1: Comparison: Brimonidine Tartrate 0.5% Gel vs Vehicle; This analysis was performed for Mobility; Test type: Superiority; p = 0.5821, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Brimonidine Tartrate 0.5% Gel vs Vehicle; This analysis was performed for Self-Care; Test type: Superiority; p = 0.8864, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Brimonidine Tartrate 0.5% Gel vs Vehicle; This analysis was performed for usual activities; Test type: Superiority; p = 0.9579, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Brimonidine Tartrate 0.5% Gel vs Vehicle; This analysis was performed for Pain/Discomfort; Test type: Superiority; p = 0.1344, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Brimonidine Tartrate 0.5% Gel vs Vehicle; Anxiety/Depression; Test type: Superiority; p = 0.1881, Cochran-Mantel-Haenszel

4. Primary Outcome: Percent Change From Baseline in Total Score of Dermatology Life Quality Index (DLQI) Questionnaire at Day 8
Description: DLQI was a compact health-related quality of life index that has 10 questions and depends on the participants self-declaration about experiences during the previous week. DLQI results range between grades 0 and 30. [Grade 0-1]: No effect at all on participant's life, [Grade 2-5]: Small effect at all on participant's life, [Grade 6-10]: Moderate effect at all on participant's life, [Grade 11-20]: Very large effect at all on participant's life, [Grade 21-30]: Extremely large effect at all on participant's life. As the DLQI scores increase, the impact of the studied disease on life becomes greater.
Time Frame: Baseline, Day 8
Population: ITT population consisted of the entire population enrolled and randomized. Here the over all number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Brimonidine Tartrate 0.5% Gel | Vehicle
Number analyzed (Participants) | 45 | 41
percent change | -15.4 (61.7) | -32.6 (43.7)
Statistical Analysis 1: Comparison: Brimonidine Tartrate 0.5% Gel vs Vehicle; Test type: Superiority; p = 0.3935, Cochran-Mantel-Haenszel

5. Primary Outcome: Euro Quality of Life-5 Dimensional-3 Level (EQ-5D-3L) Questionnaire (Along With a Visual Analogue Score for the Overall Health State) at Day 8
Description: as for outcome 3
Time Frame: Day 8
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Brimonidine Tartrate 0.5% Gel | Vehicle
Number analyzed (Participants) | 45 | 42
Score on scale | 76.0 (19.3) | 80.2 (13.1)
Statistical Analysis 1: Comparison: Brimonidine Tartrate 0.5% Gel vs Vehicle; Test type: Superiority; p = 0.4162, Cochran-Mantel-Haenszel

6. Secondary Outcome: Percentage of Participants With at Least Two Grade Improvement in the Clinician's Erythema Assessment (CEA)
Description: Evaluation of erythema by using CEA was assessed by 0 to 4 grades, where 0-Clear skin with no signs of erythema, 1- Almost clear; slight redness, 2-Mild erythema; definite redness, 3-Moderate erythema; marked redness, 4-Severe erythema; fiery redness. Percentage of participants with at least two grade improvement in the CEA was reported.
Time Frame: Day 8
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Brimonidine Tartrate 0.5% Gel | Vehicle
Number analyzed (Participants) | 46 | 42
Percentage of participants | 47.8 | 7.1

7. Secondary Outcome: Percentage of Participants With at Least Two Grade Improvement in the Participant Self-assessment
Description: Percentage of participants with at least two grade improvement in the PSA was reported. Evaluation of erythema severity by using the PSA grades (0-4): 0- No redness, 1- very mild redness, 2-mild redness, 3-moderate redness, 4-severe redness.
Time Frame: Day 8
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Brimonidine Tartrate 0.5% Gel | Vehicle
Number analyzed (Participants) | 46 | 42
Percentage of participants | 41.3 | 23.8

8. Secondary Outcome: Change From Baseline in Facial Inflammatory Lesion Counts at Day 8
Description: Facial inflammatory lesions of rosacea (including papules and pustules) were counted by evaluator.
Time Frame: Day 8
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: number of lesions
Arm/Group | Brimonidine Tartrate 0.5% Gel | Vehicle
Number analyzed (Participants) | 46 | 42
number of lesions | 0.3 (2.5) | 0.4 (1.4)

9. Secondary Outcome: Number of Participants Reported Adverse Events
Description: All clinical medical events, whether observed by the investigator or reported by the participant and whether or not thought to be product- or study procedure-related were considered as adverse events.
Time Frame: From start of study drug administration up to Day 8
Population: All Patient Treated (APT) population included all participants enrolled in the study who had received the study treatment at least once.
Measure: Count of Participants; unit: Participants
Arm/Group | Brimonidine Tartrate 0.5% Gel | Vehicle
Number analyzed (Participants) | 48 | 44
Participants | 15 | 9

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to Day 8
Arm/Group | Brimonidine Tartrate 0.5% Gel | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/44
Other Adverse Events (participants affected / at risk) | 15/48 | 9/44
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brimonidine Tartrate 0.5% Gel (N=48) | Vehicle (N=44)
Rash pustular (Infections and infestations) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 6 (6) | 2 (2)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rosacea (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin tightness (Skin and subcutaneous tissue disorders) | 4 (5) | 2 (3)
Skin warm (Skin and subcutaneous tissue disorders) | 2 (9) | 1 (2)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 2 (2) | 0 (0)
Hypoesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure agreement covered by contract.